CLINICAL TRIAL: NCT00161044
Title: An Open-Label Investigation of the Adjuvant Therapeutic Effects of Galantamine in Patients With Chronic Schizophrenia and Persistent Deficit Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, MPRC, PI, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-23059
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Chronic Schizophrenia
MeSH Terms: interventions — Galantamine

INTERVENTIONS:
Drug: Galantamine

SUMMARY:
The purpose of this study is to see if galantamine is an effective agent for the treatment of the cognitive abnormalities, negative symptoms, and /or behavioral impairments seen in schizophrenia.

DETAILED DESCRIPTION:
In this exploratory investigation, we propose to study the adjuvant therapeutic efficacy and safety of galantamine in 20 patients with chronic schizophrenia, who are maintained on a stable regimen of antipsychotic medication for at least two weeks prior to enrollment (see Table 1 for Selection Criteria). Assessments of neuropsychological performance will be made prior to the start of galantamine therapy and at study endpoint. Upon enrollment, neuropsychological tests will be administered by the study neuropsychologist, or a trained and supervised assessment technician; in fixed order, and according to standardized testing procedures. The following tests will be administered: (1) Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) (covering (a) verbal and visual episodic memory, (b) verbal response generation and self-monitoring, (c) auditory attention and working memory, and (d) sustained attention and psychomotor speed); and (2) Grooved Pegboard Test (motor speed). RBANS administration will be counterbalanced (using Forms A and B) across subjects and assessment points to prevent order effects. Remaining assessments will be administered at baseline, after galantamine titration, and at weeks 4 and 8 of galantamine treatment. Psychiatric symptoms and behavior will be assessed using the Brief Psychiatric Rating Scale (BPRS), the Scale for the Assessment of Negative Symptoms (SANS), the Montgomery-Asberg Depression Rating Scale (MADRS); the Neuropsychiatric Inventory (NPI); the Clinical Global Impression Scale (CGI); and the Apathy Evaluation Scale (AES). Trained research nurses, psychologists and psychiatrists, will administer the symptom, behavior and functional scales with established inter-rater reliability. In this study, adverse effects will be monitored through self-reporting and observation. Vital signs will be collected on a weekly basis. Additionally, motor and movement side effects will be rated by trained research nurses, using the Extrapyramidal Symptom Rating Scale (EPRS), the Barnes Akathisia Scale (BAS); and the Abnormal Involuntary Movements Scale (AIMS). Following their initial neuropsychological assessment patients will enter a ¿three week galantamine titration phase¿ during which galantamine will be added to the stable regimen of antipsychotic medication according to the following titration schedule: 8 mg/day for the first week, followed by 16 mg/day in the second and 24 mg/day in the third week (Raskin et al., 2000). At the end of this titration phase, patients will be receiving the maximal allowable dose of galantamine (i.e., 24 mg/day) or an optimal dose (i.e., the highest tolerable dose devoid of significant side effects [e.g., 16 mg/day]). Moreover, at the end of this titration phase, patients will be administered the standard battery of rating instruments prior to entering an 8-week period of active treatment with the maximal or optimal adjuvant therapeutic dose of galantamine. During the active treatment phase, the standard battery of rating instruments will be administered at the end of the fourth and eighth week of active treatment. Patients admitted to the 364A Unit at Perry Point will have their charts reviewed to see if they meet the inclusion criteria for the study. After approval by the principal investigator the patient will be approached by a designated member of the research team for their interest in participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Fulfills DSM-IV criteria for schizophrenia.
* Unable to achieve competitive employment status within the past five years.
* Unable to live independently in the community.
* Maintained on a stable regimen of antipsychotic medication for at least two weeks prior to enrollment.

Exclusion Criteria:

* History of significant hepatic, renal, pulmonary, endocrine, active peptic ulcer disease or cardiovascular disease.
* History of seizure disorder and/or head injury.
* Co-morbid substance use/abuse disorder.
* Received an investigational medication within the previous month.
* Due to the risk of adverse effects on fetal development: women with any risk of becoming pregnant will be excluded from this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2004-09; Study Completion 2005-09

PRIMARY OUTCOMES:
This trial is an exploratory open-label trial; thus, several outcome measures are employed in order to detect possible therapeutic effects in the negative symptom domain of psychopathology

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Nelson, Pharm.D., Principal Investigator — MPRC
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States